CLINICAL TRIAL: NCT03783481
Title: Distress Reduction by Activity Tracking and Activity Enhancement by Mobile Support Group in Oncology
Acronym: DRAAGON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Il Yong Chung, Principal Investigator, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: S2018-2450-0001
Record Dates: First submitted 2018-12-17; First posted 2018-12-21 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer; Mobile Community
Keywords: Breast cancer survivors; mobile community; distress
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile community group (Experimental): join the mobile community via the smartphone application
  Interventions: Device: Mobile community
- No community group (Active Comparator)
  Interventions: Other: No Mobile community

INTERVENTIONS:
Device: Mobile community — Install an application (app) on subjects' smartphone. Subject's will join the mobile community using the application through which they can check their own and other members daily steps and communicate with each other.
  Arms: Mobile community group
Other: No Mobile community — No Mobile community
  Arms: No community group

SUMMARY:
This study aims to investigate the effect of the formation of social networks using smartphones can help increase physical activity and reduce stress in survivors after breast cancer treatment surgery.

ELIGIBILITY:
Inclusion Criteria:

* Stage 0-III breast cancer
* ECOG Performance Status 0
* Patient who underwent surgery for breast cancer
* Patients with their own smartphones and who can use smartphone apps

Exclusion Criteria:

* Breast cancer recurrence or metastasis
* Severe medical illness
* need to Adjubant Chemotherapy

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Rate of moderate to severe distress at 6 months | 6months
  Using distress thermometer collected by smartphone application based questionnaire

SECONDARY OUTCOMES:
total weekly steps at 6 months | 6months
  the total number of weekly steps collected by smartphone application

CONTACTS AND LOCATIONS:
Overall Officials: Il Yong Chung, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Korea, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jung M, Lee SB, Lee JW, Park YR, Chung H, Min YH, Park HJ, Lee M, Chung S, Son BH, Ahn SH, Chung IY. The Impact of a Mobile Support Group on Distress and Physical Activity in Breast Cancer Survivors: Randomized, Parallel-Group, Open-Label, Controlled Trial. J Med Internet Res. 2023 Aug 7;25:e47158. doi: 10.2196/47158. PMID 37549004